CLINICAL TRIAL: NCT01698983
Title: Ex Vivo Stimulation of Whole Blood as a Means to Determine Glucocorticoid Sensitivity to Mild-to-Moderate and Refractory Asthmatics
Status: Terminated | Type: Observational
Why Stopped: data not as expected
Sponsor: Jeanette Marketon, MD (Other)
Responsible Party: Sponsor-Investigator, Jeanette Marketon, MD, Assistant Professor, Ohio State University
Organization: Ohio State University (Other)
Other Study IDs: 2011H0055
Record Dates: First submitted 2012-10-01; First posted 2012-10-03 (Estimated); Last update posted 2012-10-31 (Estimated); Status verified 2012-10

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Gluococorticoids are commonly prescribed to treat a number of diseases including the majority of inflammatory diseases. Despite considerable inter-personal variability in responses to glucocorticoids between asthmatics, an insensitivity rate of about 30% and the risk of adverse side effects of glucocorticoid therapy, no assay is currently performed to determine sensitivity in severe and non-severe asthmatics prior to treatment. The purpose of this study is to perform a whole blood ex vivo stimulation assay to interrogate known glucocorticoid receptor (GR) up- and down-regulated genes to indicate glucocorticoid sensitivity and compare the results between severe and non-severe asthmatics.

ELIGIBILITY:
Inclusion criteria:

To be eligible for the study, subjects must meet all of the following criteria:

* Age ≥ 18 years old
* Physician diagnosis of asthma confirmed through medical record documentation.
* Documented history of 12% FEV1 reversibility post-bronchodilator and/or Methacholine PC 20 score of 16mg/ml or less.
* Non-smoker for > 6 months before enrollment into the trial
* Less than 5 pack year smoking history defined as the average packs smoked per day multiplied by the years of active smoking.
* Willing and able to adhere to the study visit schedule and other protocol-specified procedures.

Exclusion criteria:

Subjects meeting any of the following criteria may not be enrolled in the study:

* Existence of lung disease (other than asthma)
* Recent asthma exacerbation requiring hospital admissions, unexpected healthcare visits, or prednisone courses in the previous 4 weeks.
* Non-English speaking.
* Participation in another interventional research trial
* Self-reported pregnancy
* Inability or unwillingness to provide consent
* Febrile illness (>38.0˚ C or 100.4˚ F) within 24 hours of visit.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: clinic
Sampling Method: Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2011-06; Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeanette Marketon, Ph.D., Principal Investigator — Recruit and Consent Patients
Locations (1):
- Martha Morehouse Medical Pavillion, Columbus, Ohio, United States